CLINICAL TRIAL: NCT04801420
Title: SAFETY AND IMMUNOGENICITY STUDY OF VLA15, A MULTIVALENT RECOMBINANT OSPA BASED VACCINE CANDIDATE AGAINST LYME BORRELIOSIS: A RANDOMIZED, CONTROLLED, OBSERVER-BLIND PHASE 2 STUDY IN A HEALTHY PEDIATRIC AND ADULT STUDY POPULATION
Brief Title: Phase 2 Study Of VLA15, A Vaccine Candidate Against Lyme Borreliosis, In A Healthy Pediatric And Adult Study Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VLA15-221; C4601008 (Other: Alias Study Number)
Record Dates: First submitted 2021-03-08; First posted 2021-03-17 (Actual); Results first posted 2023-06-07 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Lyme Borreliosis
Keywords: VLA15; Lyme Borreliosis; Vaccine; Lyme disease; Borrelia
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A+B - Group 1 (Experimental): Part A: VLA15 at Month 0, 2 and 6 Part B: VLA15 at Month 18, 30 and 42
  Interventions: Biological: VLA15
- Part A+B - Group 2 (Experimental): Part A: VLA15 at Month 0 and 6, placebo at Month 2 Part B: VLA15 at Month 18, 30 and 42
  Interventions: Biological: VLA15; Biological: Placebo
- Part A+B - Group 3 (Placebo Comparator): Part A: Placebo at Month 0, 2 and 6 Part B: Placebo at Month 18, 30 and 42
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VLA15 — a multivalent recombinant Outer Surface Protein A (OspA) based vaccine candidate
  Arms: Part A+B - Group 1; Part A+B - Group 2
Biological: Placebo — PBS (Phosphate Buffered Saline)
  Arms: Part A+B - Group 2; Part A+B - Group 3

SUMMARY:
VLA15-221 is a Phase 2 study, which will be conducted in two parts: Main Study Phase (Part A) and Booster Phase (Part B). The study will compare the safety and immunogenicity of two different primary immunization schedules applying three (Month 0-2-6) or two (Month 0- 6) vaccinations. Within the study, 600 healthy subjects aged 5-65 years will be included. Subjects with a history of Lyme borreliosis (previous infection with Borrelia) as well as Borrelia naïve subjects will be enrolled. Study duration per subject will be a maximum of 50 months per subject.

DETAILED DESCRIPTION:
VLA15-221 is a randomized, observer-blind, placebo controlled, multicenter Phase 2 study, which is set up in two parts: Main Study Phase (Part A) and Booster Phase (Part B). In Part A 600 subjects aged 5-65 years will be enrolled 1:1:1 into three groups: Group 1 will be vaccinated with VLA15 at Month 0-2-6, Group 2 will be vaccinated with VLA15 at Month 0-6 and with placebo at Month 2 and Group 3 will be vaccinated with placebo at Month 0-2-6. In Part B all eligible subjects will receive booster injections with VLA15 or placebo at Month 18, 30 and 42.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged 5 to 65 years at the day of screening (Visit 0)
* Subject is of good general health
* Parent(s)/legal representative(s) and subject understand the study and its procedures, agree to its provisions

  * for subjects aged 18-65 years: written informed consent prior to any study related procedures
  * for subjects aged 5-17 years: written informed consent by the subject's legal representative(s), according to local requirements, and written informed assent of the subject, if applicable, prior to any study related procedures.
* If subject is of childbearing potential: Subject has a negative serum pregnancy test at screening (Visit 0) and agrees to employ adequate birth control measures according to following timelines:

  * Main Study Phase: duration of entire study
  * Booster Phase: until 5 months after each booster vaccination (Booster 1 until Month 23, Booster 2 until Month 35 and Booster 3 until Month 47)
* Subject is willing and able to comply with scheduled visits, treatment plan, and other study procedures
* Subject is available for the duration of the study and can be contacted by telephone during study participation

Exclusion Criteria:

* Subject has a chronic illness related to Lyme borreliosis (LB), an active symptomatic LB, or received treatment for LB within the last 3 months prior to Day 1;
* Subject received previous vaccination against LB;
* Subject had a tick bite within 4 weeks prior to Day 1;
* Subject has a medical history of or currently has a clinically relevant disease;
* Subject has a medical history of or currently has a neuro- inflammatory or autoimmune disease;
* Subject has a known thrombocytopenia, bleeding disorder, or received anticoagulants in the 3 weeks prior to Day 1;
* Subject has received an active or passive immunization within 4 weeks prior to Day 1;
* Subject has received any other registered or non-registered medicinal product in another clinical trial within 4 weeks prior to vaccination at Day 1;
* Subject has a known or suspected defect of the immune system or received immuno-suppressive therapy within 4 weeks prior to Day 1;
* Subject has a history of anaphylaxis of unknown cause or severe allergic reactions of unknown cause or has a known hypersensitivity or allergic reactions to one of the components of the vaccine;
* Subject had any malignancy in the past 5 years;
* Subject is pregnant, has plans to become pregnant during the course of the study or is lactating at the time of enrollment;
* Subject has donated or plans to donate blood or blood-derived products 4 weeks prior to Day 1;
* Subject has any condition that may compromise its well-being, might interfere with evaluation of study endpoints, or would limit the subject's ability to complete the study;
* Subject is in a dependent relationship with the sponsor/investigator

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2025-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (21):
  - New England Research Associates, Bridgeport, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Pediatric Associates of Conn. PC, Waterbury, Connecticut
  - Quest Diagnostics, Marlborough, Massachusetts
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Foundation Pediatrics, East Orange, New Jersey
  - Med Clinical Research Partners, LLC, Irvington, New Jersey
  - Meridian Clinical Research LLC, Binghamton, New York
  - Pfizer Vaccine Research and Development, Pearl River, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Advantage Clinical Trials, The Bronx, New York
  - Velocity Clinical Research, Inc., Cleveland, Ohio
  - Allegheny Health and Wellness Pavilion, Erie, Pennsylvania
  - Liberty Family Practice, Erie, Pennsylvania
  - Lockman & Lubell Pediatric Associates, Fort Washington, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Velocity Clinical Research Providence, Warwick, Rhode Island
- Synevo Studien Service Labor GmbH c/o Institut für Medizinische Diagnostik, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Wagner L, Obersriebnig M, Hochreiter R, Kadlecek V, Larcher-Senn J, Hegele L, Maguire JD, Murphy T, Derhaschnig U, Bezay N, Jaramillo JC, Eder-Lingelbach S, Messier M. Immunogenicity and safety of an 18-month booster dose of the VLA15 Lyme borreliosis vaccine candidate after primary immunisation in children, adolescents, and adults in the USA: a randomised, observer-blind, placebo-controlled, phase 2 trial. Lancet Infect Dis. 2025 Nov 7:S1473-3099(25)00541-9. doi: 10.1016/S1473-3099(25)00541-9. Online ahead of print. PMID 41213278
- [Derived] Wagner L, Obersriebnig M, Kadlecek V, Hochreiter R, Ghadge SK, Larcher-Senn J, Hegele L, Maguire JD, Derhaschnig U, Jaramillo JC, Eder-Lingelbach S, Bezay N. Immunogenicity and safety of different immunisation schedules of the VLA15 Lyme borreliosis vaccine candidate in adults, adolescents, and children: a randomised, observer-blind, placebo-controlled, phase 2 trial. Lancet Infect Dis. 2025 Sep;25(9):986-999. doi: 10.1016/S1473-3099(25)00092-1. Epub 2025 Apr 25. PMID 40294611
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=VLA15-221

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 714 participants were screened of which 89 failed screening and 625 participants were randomized into the study.
Groups:
- Group 1: VLA15: Participants aged 5 to 65 years received three intramuscular vaccinations of 180 microgram (mcg) VLA15 at Month 0, 2 and 6 during the Main Study Phase. Eligible participants will receive booster dose of VLA15 at Month 18, 30 and 42 during the Booster Phase.
- Group 2: VLA15 + Placebo: Participants aged 5 to 65 years received two intramuscular vaccinations of 180 mcg VLA15 at Month 0 and 6 and a placebo injection at Month 2 during the Main Study Phase. Eligible participants will receive booster dose of VLA15 at Month 18, 30 and 42 during the Booster Phase.
- Group 3: Placebo: Participants aged 5 to 65 years received three intramuscular vaccinations of placebo at Month 0, 2 and 6 during the Main Study Phase. Eligible participants will receive placebo injection at Month 18, 30 and 42 during the Booster Phase.
Period: Overall Study
Arm/Group | Group 1: VLA15 | Group 2: VLA15 + Placebo | Group 3: Placebo
Started | 208 | 209 | 208
Completed | 0 | 0 | 0
Not Completed | 208 | 209 | 208
Not completed — Other | 1 | 2 | 1
Not completed — Lost to Follow-up | 7 | 9 | 10
Not completed — Moved from study area | 0 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 1 | 4
Not completed — Individual stopping criteria reached | 0 | 1 | 0
Not completed — Ongoing in the study | 195 | 195 | 192

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all participants enrolled who received at least one vaccination. Participants were analyzed according to the study group they were allocated to, rather than by the actual treatment they received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: VLA15 | Group 2: VLA15 + Placebo | Group 3: Placebo | Total
Number analyzed (Participants) | 208 | 209 | 208 | 625
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.7 (19.08) | 28.9 (19.56) | 29.0 (19.72) | 28.9 (19.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 108 | 101 | 321
  Male | 96 | 101 | 107 | 304
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 4 | 3 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 27 | 17 | 24 | 68
  White | 172 | 184 | 176 | 532
  Unknown or Not Reported | 4 | 5 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Local and Solicited Systemic Adverse Events (AEs) Within 7 Days After Vaccination 1
Description: Participants or their legal guardians were required to record any solicited local and systemic adverse events in the electronic diary. Solicited symptoms were pre-defined symptoms which were collected via an electronic diary. Solicited local AEs included pain, tenderness, erythema (redness), swelling and induration (hardening). Solicited systemic AEs included headache, muscle pain, joint pain, nausea, vomiting, fatigue and fever. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: From Day 1 to Day 7 after vaccination 1 at Month 0
Population: Safety Analysis Set (SAS) included all participants who entered into the study and received at least one vaccination. Participants were analyzed according to the actual treatment received. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Any VLA15: Participants aged 5 to 65 years who received intramuscular vaccinations of 180 mcg VLA15 at either Month 0, 2 or 6 during the Main Study Phase were included. This arm also included participants who received wrong vaccination or missed a vaccination and could not be assigned to Group 1 or 2.
- All Participants: Participants aged 5 to 65 years who received intramuscular vaccination of either 180 mcg VLA15 or placebo during the Main Study Phase were included. This arm also included participants who received wrong vaccination or missed a vaccination.
Arm/Group | Group 1: VLA15 | Group 2: VLA15 + Placebo | Group 3: Placebo | Any VLA15 | All Participants
Number analyzed (Participants) | 190 | 187 | 208 | 417 | 625
Percentage of participants
  Pain: number analyzed (Participants) | 184 | 182 | 200 | 402 | 602
  Pain | 63.0 [55.9 to 69.7] | 59.3 [52.1 to 66.2] | 12.5 [8.6 to 17.8] | 60.4 [55.6 to 65.1] | 44.5 [40.6 to 48.5]
  Tenderness: number analyzed (Participants) | 185 | 184 | 200 | 406 | 606
  Tenderness | 81.6 [75.4 to 86.5] | 84.8 [78.9 to 89.3] | 19.5 [14.6 to 25.5] | 81.8 [77.7 to 85.2] | 61.2 [57.3 to 65.0]
  Erythema/redness: number analyzed (Participants) | 181 | 181 | 199 | 397 | 596
  Erythema/redness | 12.2 [8.2 to 17.7] | 14.9 [10.5 to 20.8] | 2.5 [1.1 to 5.7] | 13.1 [10.1 to 16.8] | 9.6 [7.5 to 12.2]
  Swelling: number analyzed (Participants) | 179 | 181 | 200 | 394 | 594
  Swelling | 8.9 [5.6 to 14.0] | 8.8 [5.5 to 13.9] | 0.5 [0.1 to 2.8] | 9.1 [6.7 to 12.4] | 6.2 [4.6 to 8.5]
  Induration/Hardening: number analyzed (Participants) | 180 | 181 | 199 | 395 | 594
  Induration/Hardening | 10.0 [6.4 to 15.3] | 6.6 [3.8 to 11.2] | 1.0 [0.3 to 3.6] | 8.9 [6.4 to 12.1] | 6.2 [4.6 to 8.5]
  Headache: number analyzed (Participants) | 181 | 180 | 200 | 396 | 596
  Headache | 24.9 [19.1 to 31.6] | 21.1 [15.8 to 27.6] | 19.5 [14.6 to 25.5] | 23.5 [19.6 to 27.9] | 22.1 [19.0 to 25.7]
  Muscle pain: number analyzed (Participants) | 183 | 182 | 200 | 401 | 601
  Muscle pain | 36.1 [29.5 to 43.2] | 34.6 [28.1 to 41.8] | 11.0 [7.4 to 16.1] | 35.7 [31.1 to 40.5] | 27.5 [24.0 to 31.2]
  Joint pain: number analyzed (Participants) | 181 | 180 | 201 | 395 | 596
  Joint pain | 9.9 [6.4 to 15.2] | 3.9 [1.9 to 7.8] | 6.5 [3.8 to 10.7] | 7.6 [5.4 to 10.6] | 7.2 [5.4 to 9.6]
  Nausea: number analyzed (Participants) | 178 | 180 | 200 | 392 | 592
  Nausea | 3.9 [1.9 to 7.9] | 6.1 [3.4 to 10.6] | 6.0 [3.5 to 10.2] | 5.4 [3.5 to 8.1] | 5.6 [4.0 to 7.7]
  Vomiting: number analyzed (Participants) | 178 | 180 | 199 | 392 | 591
  Vomiting | 1.1 [0.3 to 4.0] | 0.6 [0.1 to 3.1] | 1.0 [0.3 to 3.6] | 0.8 [0.3 to 2.2] | 0.8 [0.4 to 2.0]
  Fatigue: number analyzed (Participants) | 179 | 181 | 201 | 395 | 596
  Fatigue | 20.7 [15.4 to 27.2] | 17.1 [12.3 to 23.3] | 16.4 [11.9 to 22.2] | 19.7 [16.1 to 24.0] | 18.6 [15.7 to 21.9]
  Fever: number analyzed (Participants) | 167 | 163 | 188 | 363 | 551
  Fever | 1.8 [0.6 to 5.1] | 0.0 [0.0 to 2.3] | 0.5 [0.1 to 3.0] | 1.1 [0.4 to 2.8] | 0.9 [0.4 to 2.1]

2. Primary Outcome: Percentage of Participants With Solicited Local and Solicited Systemic AEs Within 7 Days After Vaccination 2
Description: as for outcome 1
Time Frame: From Day 1 to Day 7 after vaccination 2 at Month 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: VLA15 | Group 2: VLA15 + Placebo | Group 3: Placebo | Any VLA15 | All Participants
Number analyzed (Participants) | 190 | 181 | 203 | 399 | 602
Percentage of participants
  Pain: number analyzed (Participants) | 185 | 177 | 191 | 390 | 581
  Pain | 56.8 [49.6 to 63.7] | 7.9 [4.8 to 12.8] | 8.4 [5.2 to 13.2] | 32.1 [27.6 to 36.8] | 24.3 [21.0 to 27.9]
  Tenderness: number analyzed (Participants) | 188 | 177 | 193 | 393 | 586
  Tenderness | 81.4 [75.2 to 86.3] | 14.7 [10.2 to 20.7] | 14.5 [10.2 to 20.2] | 47.6 [42.7 to 52.5] | 36.7 [32.9 to 40.7]
  Erythema/redness: number analyzed (Participants) | 184 | 177 | 191 | 388 | 579
  Erythema/redness | 15.8 [11.2 to 21.7] | 0.0 [0.0 to 2.1] | 1.6 [0.5 to 4.5] | 7.5 [5.3 to 10.5] | 5.5 [3.9 to 7.7]
  Swelling: number analyzed (Participants) | 184 | 177 | 191 | 387 | 578
  Swelling | 11.4 [7.6 to 16.8] | 0.0 [0.0 to 2.1] | 0.5 [0.1 to 2.9] | 5.4 [3.6 to 8.2] | 3.8 [2.5 to 5.7]
  Induration/Hardening: number analyzed (Participants) | 185 | 177 | 191 | 390 | 581
  Induration/Hardening | 9.2 [5.8 to 14.2] | 1.1 [0.3 to 4.0] | 0.0 [0.0 to 2.0] | 5.4 [3.5 to 8.1] | 3.6 [2.4 to 5.5]
  Headache: number analyzed (Participants) | 184 | 176 | 192 | 386 | 578
  Headache | 16.8 [12.1 to 22.9] | 12.5 [8.4 to 18.2] | 13.0 [9.0 to 18.5] | 15.3 [12.0 to 19.2] | 14.5 [11.9 to 17.6]
  Muscle pain: number analyzed (Participants) | 185 | 176 | 191 | 388 | 579
  Muscle pain | 23.8 [18.2 to 30.4] | 4.0 [1.9 to 8.0] | 3.7 [1.8 to 7.4] | 14.2 [11.1 to 18.0] | 10.7 [8.4 to 13.5]
  Joint pain: number analyzed (Participants) | 184 | 176 | 191 | 386 | 577
  Joint pain | 4.9 [2.6 to 9.0] | 3.4 [1.6 to 7.2] | 1.6 [0.5 to 4.5] | 4.7 [3.0 to 7.3] | 3.6 [2.4 to 5.5]
  Nausea: number analyzed (Participants) | 184 | 176 | 193 | 385 | 578
  Nausea | 4.3 [2.2 to 8.3] | 3.4 [1.6 to 7.2] | 5.7 [3.2 to 9.9] | 3.6 [2.2 to 6.0] | 4.3 [2.9 to 6.3]
  Vomiting: number analyzed (Participants) | 184 | 176 | 191 | 385 | 576
  Vomiting | 1.1 [0.3 to 3.9] | 1.7 [0.6 to 4.9] | 0.0 [0.0 to 2.0] | 1.3 [0.6 to 3.0] | 0.9 [0.4 to 2.0]
  Fatigue: number analyzed (Participants) | 184 | 176 | 192 | 385 | 577
  Fatigue | 13.6 [9.4 to 19.3] | 9.1 [5.7 to 14.3] | 12.0 [8.1 to 17.3] | 11.9 [9.1 to 15.6] | 12.0 [9.6 to 14.9]
  Fever: number analyzed (Participants) | 176 | 167 | 182 | 368 | 550
  Fever | 1.7 [0.6 to 4.9] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.1] | 0.8 [0.3 to 2.4] | 0.5 [0.2 to 1.6]

3. Primary Outcome: Percentage of Participants With Solicited Local and Solicited Systemic AEs Within 7 Days After Vaccination 3
Description: as for outcome 1
Time Frame: From Day 1 to Day 7 after vaccination 3 at Month 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: VLA15 | Group 2: VLA15 + Placebo | Group 3: Placebo | Any VLA15 | All Participants
Number analyzed (Participants) | 190 | 187 | 191 | 384 | 575
Percentage of participants
  Pain: number analyzed (Participants) | 178 | 178 | 179 | 363 | 542
  Pain | 57.3 [50.0 to 64.3] | 62.4 [55.1 to 69.1] | 5.6 [3.1 to 10.0] | 59.5 [54.4 to 64.4] | 41.7 [37.6 to 45.9]
  Tenderness: number analyzed (Participants) | 179 | 179 | 179 | 365 | 544
  Tenderness | 74.3 [67.4 to 80.1] | 83.2 [77.1 to 88.0] | 12.8 [8.7 to 18.5] | 78.6 [74.1 to 82.5] | 57.0 [52.8 to 61.1]
  Erythema/redness: number analyzed (Participants) | 178 | 177 | 179 | 362 | 541
  Erythema/redness | 10.7 [6.9 to 16.1] | 7.9 [4.8 to 12.8] | 1.1 [0.3 to 4.0] | 9.7 [7.0 to 13.1] | 6.8 [5.0 to 9.3]
  Swelling: number analyzed (Participants) | 177 | 177 | 179 | 361 | 540
  Swelling | 7.9 [4.8 to 12.8] | 10.2 [6.5 to 15.5] | 0.6 [0.1 to 3.1] | 9.1 [6.6 to 12.6] | 6.3 [4.5 to 8.7]
  Induration/Hardening: number analyzed (Participants) | 177 | 178 | 179 | 362 | 541
  Induration/Hardening | 7.9 [4.8 to 12.8] | 9.0 [5.6 to 14.1] | 0.6 [0.1 to 3.1] | 8.3 [5.9 to 11.6] | 5.7 [4.1 to 8.0]
  Headache: number analyzed (Participants) | 175 | 178 | 180 | 360 | 540
  Headache | 16.6 [11.8 to 22.8] | 20.8 [15.5 to 27.3] | 8.9 [5.5 to 14.0] | 18.6 [14.9 to 23.0] | 15.4 [12.6 to 18.7]
  Muscle pain: number analyzed (Participants) | 176 | 179 | 179 | 362 | 541
  Muscle pain | 26.7 [20.7 to 33.7] | 29.6 [23.4 to 36.7] | 7.8 [4.7 to 12.7] | 28.2 [23.8 to 33.0] | 21.4 [18.2 to 25.1]
  Joint pain: number analyzed (Participants) | 175 | 178 | 180 | 360 | 540
  Joint pain | 6.3 [3.5 to 10.9] | 3.9 [1.9 to 7.9] | 3.3 [1.5 to 7.1] | 5.0 [3.2 to 7.8] | 4.4 [3.0 to 6.5]
  Nausea: number analyzed (Participants) | 175 | 177 | 179 | 359 | 538
  Nausea | 2.3 [0.9 to 5.7] | 4.0 [1.9 to 7.9] | 2.2 [0.9 to 5.6] | 3.1 [1.7 to 5.4] | 2.8 [1.7 to 4.5]
  Vomiting: number analyzed (Participants) | 175 | 177 | 179 | 359 | 538
  Vomiting | 1.1 [0.3 to 4.1] | 1.1 [0.3 to 4.0] | 0.0 [0.0 to 2.1] | 1.1 [0.4 to 2.8] | 0.7 [0.3 to 1.9]
  Fatigue: number analyzed (Participants) | 175 | 178 | 180 | 360 | 540
  Fatigue | 17.7 [12.8 to 24.0] | 16.9 [12.1 to 23.0] | 11.7 [7.8 to 17.2] | 17.2 [13.7 to 21.5] | 15.4 [12.6 to 18.7]
  Fever: number analyzed (Participants) | 169 | 170 | 173 | 346 | 519
  Fever | 0.0 [0.0 to 2.2] | 1.8 [0.6 to 5.1] | 0.6 [0.1 to 3.2] | 0.9 [0.3 to 2.5] | 0.8 [0.3 to 2.0]

4. Primary Outcome: Percentage of Participants With Solicited Local and Solicited Systemic AEs Within 7 Days After Any Vaccination During the Main Study Phase
Description: as for outcome 1
Time Frame: From Day 1 to Day 7 after vaccination 1, 2 or 3 at Month 0, 2 and 6 respectively
Population: Safety Analysis Set (SAS) included all participants who entered into the study and received at least one vaccination. Participants were analyzed according to the actual treatment received. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table and for each specified row.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: VLA15 | Group 2: VLA15 + Placebo | Group 3: Placebo | Any VLA15 | All Participants
Number analyzed (Participants) | 190 | 187 | 208 | 417 | 625
Percentage of participants
  Pain | 80.5 [74.3 to 85.5] | 77.0 [70.5 to 82.5] | 16.8 [12.4 to 22.5] | 77.0 [72.7 to 80.8] | 57.0 [53.0 to 60.8]
  Tenderness | 92.6 [88.0 to 95.6] | 92.5 [87.8 to 95.5] | 28.4 [22.7 to 34.8] | 90.6 [87.5 to 93.1] | 69.9 [66.2 to 73.4]
  Erythema/Redness | 26.8 [21.0 to 33.6] | 18.7 [13.8 to 24.9] | 3.4 [1.6 to 6.8] | 21.8 [18.1 to 26.0] | 15.7 [13.0 to 18.7]
  Swelling | 20.5 [15.4 to 26.8] | 16.6 [11.9 to 22.6] | 1.4 [0.5 to 4.2] | 18.0 [14.6 to 22.0] | 12.5 [10.1 to 15.3]
  Induration/Hardening | 19.5 [14.5 to 25.7] | 14.4 [10.1 to 20.2] | 1.4 [0.5 to 4.2] | 16.5 [13.3 to 20.4] | 11.5 [9.2 to 14.3]
  Headache | 38.4 [31.8 to 45.5] | 36.4 [29.8 to 43.5] | 28.8 [23.1 to 35.3] | 37.4 [32.9 to 42.1] | 34.6 [30.9 to 38.4]
  Muscle pain | 45.8 [38.9 to 52.9] | 48.1 [41.1 to 55.3] | 17.8 [13.2 to 23.6] | 46.8 [42.0 to 51.6] | 37.1 [33.4 to 41.0]
  Joint pain | 15.3 [10.8 to 21.1] | 9.6 [6.2 to 14.7] | 8.2 [5.2 to 12.7] | 13.2 [10.3 to 16.8] | 11.5 [9.2 to 14.3]
  Nausea | 8.4 [5.2 to 13.2] | 11.2 [7.5 to 16.6] | 9.6 [6.3 to 14.4] | 9.6 [7.1 to 12.8] | 9.6 [7.5 to 12.2]
  Vomiting | 3.2 [1.5 to 6.7] | 3.2 [1.5 to 6.8] | 1.0 [0.3 to 3.4] | 2.9 [1.7 to 5.0] | 2.2 [1.3 to 3.7]
  Fatigue | 33.2 [26.9 to 40.1] | 29.9 [23.8 to 36.9] | 28.4 [22.7 to 34.8] | 31.4 [27.1 to 36.0] | 30.4 [26.9 to 34.1]
  Fever | 3.2 [1.5 to 6.7] | 1.6 [0.5 to 4.6] | 1.0 [0.3 to 3.4] | 2.4 [1.3 to 4.4] | 1.9 [1.1 to 3.3]

5. Primary Outcome: Geometric Mean Titers (GMTs) for Immunoglobulin G (IgG) Against Each Outer Surface Protein A (OspA) Serotype (ST1 to ST6) at Day 208 During the Main Study Phase
Description: GMTs for IgG against each OspA serotype ST1 to ST6, determined by an IgG binding assay at Day 208 is presented in this outcome measure.
Time Frame: Day 208 (Month 7)
Population: Per-Protocol Analysis Set (PPAS) consisted of the FAS population excluding those participants with at least one relevant protocol deviation (i.e., a protocol deviation with possible impact on immunogenicity). All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, "Number Analyzed" signifies participants with available results for each serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Units per milliliter
Arm/Group | Group 1: VLA15 | Group 2: VLA15 + Placebo | Group 3: Placebo
Number analyzed (Participants) | 177 | 162 | 177
Units per milliliter
  ST1: number analyzed (Participants) | 172 | 158 | 166
  ST1 | 333.2 [275.2 to 403.4] | 197.3 [156.2 to 249.3] | 23.8 [21.6 to 26.2]
  ST2: number analyzed (Participants) | 172 | 158 | 166
  ST2 | 656.0 [560.2 to 768.2] | 460.3 [370.6 to 571.8] | 21.9 [20.2 to 23.7]
  ST3: number analyzed (Participants) | 172 | 158 | 166
  ST3 | 586.4 [497.4 to 691.4] | 436.2 [344.8 to 551.8] | 21.9 [20.2 to 23.8]
  ST4: number analyzed (Participants) | 172 | 158 | 166
  ST4 | 422.8 [355.3 to 503.1] | 245.8 [196.1 to 308.2] | 23.5 [21.3 to 25.8]
  ST5: number analyzed (Participants) | 172 | 158 | 166
  ST5 | 443.4 [375.5 to 523.6] | 239.4 [190.5 to 301.0] | 22.4 [20.6 to 24.4]
  ST6: number analyzed (Participants) | 172 | 158 | 166
  ST6 | 429.7 [360.2 to 512.8] | 222.0 [177.4 to 277.8] | 24.3 [22.1 to 26.7]

6. Secondary Outcome: Percentage of Participants With Solicited Local and Solicited Systemic AEs Within 7 Days After Booster Dose
Description: Participants or their legal guardians were required to record any solicited local and systemic adverse events in the electronic diary. Solicited local AEs included pain, tenderness, erythema (redness), swelling and induration (hardening). Solicited systemic AEs included headache, muscle pain, joint pain, nausea, vomiting, fatigue and fever.
Time Frame: Within 7 days after booster dose
Reporting Status: Not Posted, anticipated posting 2027-01

7. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: SAE was any untoward medical occurrence that at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; was another medically important condition. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: From Day 1 of vaccination up to Day 208 (Month 7)
Population: Safety Analysis Set (SAS) included all participants who entered into the study and received at least one vaccination. Participants were analyzed according to the actual treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: VLA15 | Group 2: VLA15 + Placebo | Group 3: Placebo | Any VLA15 | All Participants
Number analyzed (Participants) | 190 | 187 | 208 | 417 | 625
Percentage of participants | 0.0 [0.0 to 2.0] | 1.1 [0.3 to 3.8] | 1.9 [0.8 to 4.8] | 0.7 [0.2 to 2.1] | 1.1 [0.5 to 2.3]

8. Secondary Outcome: Percentage of Participants With Adverse Events of Special Interest (AESIs)
Description: An AESI (serious or non-serious) was one of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor were appropriate. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: From Day 1 of vaccination up to Day 208 (Month 7)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: VLA15 | Group 2: VLA15 + Placebo | Group 3: Placebo | Any VLA15 | All Participants
Number analyzed (Participants) | 190 | 187 | 208 | 417 | 625
Percentage of participants | 0.0 [0.0 to 2.0] | 0.5 [0.1 to 3.0] | 0.0 [0.0 to 1.8] | 1.2 [0.5 to 2.8] | 0.8 [0.3 to 1.9]

9. Secondary Outcome: Percentage of Participants With Unsolicited Adverse Events
Description: An AE was any untoward medical occurrence in a participant administered an investigational product, whether or not related to this treatment. Unsolicited AEs were defined as any solicited local or systemic AE if it had an onset date more than 6 days after vaccination or any other symptom or untoward medical event. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: From Day 1 to Day 28 after vaccination 1, 2 and 3 at Month 0, 2 and 6, respectively
Population: Safety Analysis Set (SAS) included all participants who entered into the study and received at least one vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: VLA15 | Group 2: VLA15 + Placebo | Group 3: Placebo | Any VLA15 | All Participants
Number analyzed (Participants) | 190 | 187 | 208 | 417 | 625
Percentage of participants | 16.8 [12.2 to 22.8] | 25.1 [19.5 to 31.8] | 24.5 [19.2 to 30.8] | 20.9 [17.2 to 25.0] | 22.1 [19.0 to 25.5]

10. Secondary Outcome: Percentage of Participants With SAEs, AESIs, Solicited and Unsolicited AEs Stratified by Age Group
Description: Percentage of participants with SAEs, AESIs, solicited and unsolicited AEs stratified by age group 18 to 65, 12 to 17 and 5 to 11 years were reported. SAE: any untoward medical occurrence that at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; was another medically important condition. AESI: scientific and medical concern specific to the sponsor's product or program. Solicited AE: predefined reactions at injection site or systemic reactions after each vaccination. Unsolicited AEs: any solicited local or systemic AE if it had an onset date more than 6 days after vaccination or any other symptom or untoward medical event. Unsolicited AEs were collected only up to 28 days after any vaccination. Two-sided 95% confidence intervals were calculated according to Altman method.
Time Frame: SAEs, AESIs: From Day 1 of vaccination (vac) up to Day 208 (Month 7), Solicited AEs: From Day 1 to Day 7 after vac 1, 2 and 3 at Month 0, 2 and 6, respectively; Unsolicited AEs: From Day 1 to Day 28 after vac 1, 2 and 3 at Month 0, 2 and 6, respectively
Population: Safety Analysis Set (SAS) included all participants who entered into the study and received at least one vaccination. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: VLA15 | Group 2: VLA15 + Placebo | Group 3: Placebo | Any VLA15 | All Participants
Number analyzed (Participants) | 190 | 187 | 208 | 417 | 625
Percentage of participants
  SAE: 18 to 65 years: number analyzed (Participants) | 97 | 90 | 107 | 213 | 320
  SAE: 18 to 65 years | 0.0 [0.0 to 3.8] | 1.1 [0.2 to 6.0] | 1.9 [0.5 to 6.6] | 0.5 [0.1 to 2.6] | 0.9 [0.3 to 2.7]
  SAE: 12 to 17 years: number analyzed (Participants) | 44 | 48 | 50 | 100 | 150
  SAE: 12 to 17 years | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.4] | 4.0 [1.1 to 13.5] | 1.0 [0.2 to 5.4] | 2.0 [0.7 to 5.7]
  SAE: 5 to 11 years: number analyzed (Participants) | 49 | 49 | 51 | 104 | 155
  SAE: 5 to 11 years | 0.0 [0.0 to 7.3] | 2.0 [0.4 to 10.7] | 0.0 [0.0 to 7.0] | 1.0 [0.2 to 5.2] | 0.6 [0.1 to 3.6]
  AESI: 18 to 65 years: number analyzed (Participants) | 97 | 90 | 107 | 213 | 320
  AESI: 18 to 65 years | 0.0 [0.0 to 3.8] | 0.0 [0.0 to 4.1] | 0.0 [0.0 to 3.5] | 0.9 [0.3 to 3.4] | 0.6 [0.2 to 2.2]
  AESI: 12 to 17 years: number analyzed (Participants) | 44 | 48 | 50 | 100 | 150
  AESI: 12 to 17 years | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.1] | 1.0 [0.2 to 5.4] | 0.7 [0.1 to 3.7]
  AESI: 5 to 11 years: number analyzed (Participants) | 49 | 49 | 51 | 104 | 155
  AESI: 5 to 11 years | 0.0 [0.0 to 7.3] | 2.0 [0.4 to 10.7] | 0.0 [0.0 to 7.0] | 1.9 [0.5 to 6.7] | 1.3 [0.4 to 4.6]
  Solicited AE: 18 to 65 years: number analyzed (Participants) | 97 | 90 | 107 | 213 | 320
  Solicited AE: 18 to 65 years | 94.8 [88.5 to 97.8] | 95.6 [89.1 to 98.3] | 62.6 [53.2 to 71.2] | 93.9 [89.8 to 96.4] | 83.4 [79.0 to 87.1]
  Solicited AE: 12 to 17 years: number analyzed (Participants) | 44 | 48 | 50 | 100 | 150
  Solicited AE: 12 to 17 years | 97.7 [88.2 to 99.6] | 93.8 [83.2 to 97.9] | 60.0 [46.2 to 72.4] | 95.0 [88.8 to 97.8] | 83.3 [76.6 to 88.4]
  Solicited AE: 5 to 11 years: number analyzed (Participants) | 49 | 49 | 51 | 104 | 155
  Solicited AE: 5 to 11 years | 87.8 [75.8 to 94.3] | 98.0 [89.3 to 99.6] | 64.7 [51.0 to 76.4] | 93.3 [86.8 to 96.7] | 83.9 [77.3 to 88.8]
  Unsolicited AE: 18 to 65 years: number analyzed (Participants) | 97 | 90 | 107 | 213 | 320
  Unsolicited AE: 18 to 65 years | 23.7 [16.4 to 33.1] | 30.0 [21.5 to 40.1] | 29.0 [21.2 to 38.2] | 26.3 [20.8 to 32.6] | 27.2 [22.6 to 32.3]
  Unsolicited AE: 12 to 17 years: number analyzed (Participants) | 44 | 48 | 50 | 100 | 150
  Unsolicited AE: 12 to 17 years | 18.2 [9.5 to 32.0] | 20.8 [11.7 to 34.3] | 22.0 [12.8 to 35.2] | 19.0 [12.5 to 27.8] | 20.0 [14.4 to 27.1]
  Unsolicited AE: 5 to 11 years: number analyzed (Participants) | 49 | 49 | 51 | 104 | 155
  Unsolicited AE: 5 to 11 years | 2.0 [0.4 to 10.7] | 20.4 [11.5 to 33.6] | 17.6 [9.6 to 30.3] | 11.5 [6.7 to 19.1] | 13.5 [9.0 to 19.8]

11. Secondary Outcome: GMTs for IgG Against Each OspA Serotype (ST1 to ST6) at Baseline, Day 85, Day 180 and Day 194 During the Main Study Phase
Description: GMTs for IgG against each OspA serotype ST1 to ST6, determined by an IgG binding assay.
Time Frame: Baseline, Day 85, Day 180 and Day 194
Reporting Status: Not Posted, anticipated posting 2027-01

12. Secondary Outcome: Seroconversion Rate for Each OspA Serotype (ST1 to ST6) Specific IgG at Day 85, 180, 194 and 208
Description: Seroconversion Rate (SCR) for each OspA serotype specific IgG ST1 to ST6, determined by enzyme linked immunosorbent assay (ELISA). Seroconversion for ELISA was defined as: 1) For participants who were seronegative at screening: percentage of participants with a change from seronegative at screening to seropositive (i.e. antibody titer of >=40 Units per milliliter [U/mL]) at a certain time point. 2) For participants who were seropositive at screening: percentage of participants with a >= 4-fold rise in OspA IgG antibody titer from screening.
Time Frame: Day 85, Day 180, Day 194 and Day 208
Reporting Status: Not Posted, anticipated posting 2027-01

13. Secondary Outcome: Geometric Mean of the Fold Rise (GMFR) for IgG Against Each OspA Serotype (ST1 to ST6) at Day 85 and Day 208 During the Main Study Phase
Description: GMFR as compared to baseline for IgG against each OspA serotype ST1 to ST6, determined by IgG binding assay at Day 85 and Day 208.
Time Frame: Baseline, Day 85 and 208
Reporting Status: Not Posted, anticipated posting 2027-01

14. Secondary Outcome: GMTs for IgG Against Each OspA Serotype (ST1 to ST6) Stratified by Age Group at Baseline, Day 85, Day 180, Day 194 and Day 208 During the Main Study Phase
Description: GMTs for IgG against each OspA serotype ST1 to ST6, determined by an IgG binding assay stratified by age group (18 to 65, 12 to 17 and 5 to 11 years).
Time Frame: Baseline, Day 85, Day 180, Day 194 (18 to 65 years only) and Day 208
Reporting Status: Not Posted, anticipated posting 2027-01

15. Secondary Outcome: Seroconversion Rate for Each OspA Serotype (ST1 to ST6) Specific IgG at Day 85, 180, 194 and 208 Stratified by Age Group During the Main Study Phase
Description: SCR for each OspA serotype specific IgG ST1 to ST6, determined by ELISA stratified by age group (18 to 65, 12 to 17 and 5 to 11 years). Seroconversion for ELISA was defined as: 1) For participants who were seronegative at screening: percentage of participants with a change from seronegative at screening to seropositive (i.e. antibody titer of >=40 Units per milliliter [U/mL]) at a certain time point. 2) For participants who were seropositive at screening: percentage of participants with a >= 4-fold rise in OspA IgG antibody titer from screening.
Time Frame: Day 85, Day 180, Day 194 (18 to 65 years only) and Day 208
Reporting Status: Not Posted, anticipated posting 2027-01

16. Secondary Outcome: Geometric Mean of the Fold Rise (GMFR) for IgG Against Each OspA Serotype (ST1 to ST6) at Day 85, Day 180, Day 194 and Day 208 Stratified by Age Group During the Main Study Phase
Description: GMFR as compared to baseline for IgG against each OspA serotype ST1 to ST6, stratified by age group (18 to 65, 12 to 17 and 5 to 11 years) determined by IgG binding assay at Day 85, Day 180, Day 194 (18 to 65 years only) and Day 208.
Time Frame: Baseline, Day 85, Day 180, Day 194 (18 to 65 years only) and Day 208
Reporting Status: Not Posted, anticipated posting 2027-01

17. Secondary Outcome: GMTs for IgG Against Each OspA Serotype (ST1 to ST6) During the Booster Phase
Time Frame: Up to Month 48
Reporting Status: Not Posted, anticipated posting 2027-01

18. Secondary Outcome: SCR for Each OspA Serotype (ST1 to ST6) IgG During the Booster Phase
Description: Seroconversion for ELISA was defined as: 1) For participants who were seronegative at screening: a change from seronegative at screening to seropositive (i.e. antibody titer of >=40 U/mL) at a certain time point. 2) For participants who were seropositive at screening: a >= 4-fold rise in OspA IgG antibody titer from screening.
Time Frame: Up to Month 48
Reporting Status: Not Posted, anticipated posting 2027-01

19. Secondary Outcome: GMFR for IgG Against Each OspA Serotype (ST1 to ST6) at Month 19 During the Booster Phase
Time Frame: Month 19
Reporting Status: Not Posted, anticipated posting 2027-01

20. Secondary Outcome: GMTs for IgG Against Each OspA Serotype (ST1 to ST6) Stratified by Age Cohort During the Booster Phase
Time Frame: Up to Month 48
Reporting Status: Not Posted, anticipated posting 2027-01

21. Secondary Outcome: SCR for Each OspA Serotype (ST1 to ST6) IgG Stratified by Age Cohort During the Booster Phase
Description: as for outcome 18
Time Frame: Up to Month 48
Reporting Status: Not Posted, anticipated posting 2027-01

22. Secondary Outcome: GMFR for IgG Against Each OspA Serotype (ST1 to ST6) Stratified by Age Cohort During the Booster Phase
Time Frame: Up to Month 48
Reporting Status: Not Posted, anticipated posting 2027-01

ADVERSE EVENTS:
Time Frame: Solicited AEs (systematic assessment): From Day 1 to Day 7 after vaccination 1, 2 and 3 at Month 0, 2 and 6, respectively; unsolicited AEs (non-systematic assessment): From Day 1 to Day 28 after vaccination 1, 2 and 3, at Month 0, 2 and 6, respectively, all-cause mortality, AESIs and serious AEs (non-systematic assessment): From Day 1 of vaccination up to Day 208 (Month 7).
Description: Solicited AEs comprised injection site reactions (pain, tenderness, erythema [redness]), induration [hardening], swelling, or systemic reactions (headache, muscle pain, joint pain, fever, nausea, vomiting, fatigue). Solicited AEs were collected by systematic assessment through participant e-diaries. Safety Analysis Set: participants who entered into study and received at least 1 dose of vaccination. Participants were analyzed according to the actual treatment received.
Arm/Group | Group 1: VLA15 | Group 2: VLA15 + Placebo | Group 3: Placebo | Any VLA15 | All Participants
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/187 | 0/208 | 0/417 | 0/625
Serious Adverse Events (participants affected / at risk) | 0/190 | 2/187 | 4/208 | 3/417 | 7/625
Other Adverse Events (participants affected / at risk) | 178/190 | 179/187 | 133/208 | 391/417 | 524/625
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: VLA15 (N=190) | Group 2: VLA15 + Placebo (N=187) | Group 3: Placebo (N=208) | Any VLA15 (N=417) | All Participants (N=625)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Reactive attachment disorder of infancy or early childhood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: VLA15 (N=190) | Group 2: VLA15 + Placebo (N=187) | Group 3: Placebo (N=208) | Any VLA15 (N=417) | All Participants (N=625)
Injection site pain (General disorders) | 177 (760) | 176 (561) | 67 (141) | 384 (1385) | 451 (1526)
Fatigue (General disorders) | 63 (93) | 55 (77) | 59 (78) | 129 (186) | 188 (264)
Injection site erythema (General disorders) | 74 (118) | 62 (86) | 18 (23) | 147 (215) | 165 (238)
Injection site swelling (General disorders) | 64 (89) | 55 (67) | 13 (14) | 125 (162) | 138 (176)
Injection site induration (General disorders) | 56 (86) | 50 (61) | 10 (12) | 113 (158) | 123 (170)
Myalgia (Musculoskeletal and connective tissue disorders) | 87 (158) | 90 (122) | 37 (43) | 195 (300) | 232 (343)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (38) | 19 (22) | 18 (23) | 57 (71) | 75 (94)
Headache (Nervous system disorders) | 74 (106) | 68 (98) | 63 (83) | 157 (220) | 220 (303)
Nausea (Gastrointestinal disorders) | 16 (19) | 21 (25) | 20 (27) | 40 (47) | 60 (74)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/20/NCT04801420/Prot_002.pdf
  • Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT04801420/SAP_001.pdf